CLINICAL TRIAL: NCT03973034
Title: Clinical Application of ctDNA in Early Screening of Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-BREAST-ctDNA screening
Record Dates: First submitted 2019-06-02; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer
Keywords: ctDNA; early screening; Copy Number Variants (CNV); Low Depth Whole Genome Sequencing (LDWGS)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal people
  Interventions: Diagnostic Test: Low depth whole genome sequencing
- Benign breast disease patients
  Interventions: Diagnostic Test: Low depth whole genome sequencing
- Breast cancer patients in early stage
  Interventions: Diagnostic Test: Low depth whole genome sequencing

INTERVENTIONS:
Diagnostic Test: Low depth whole genome sequencing — Low depth whole genome sequencing of the peripheral blood samples from different groups.

SUMMARY:
The investigators aim to evaluate the possibility of clinical application of ctDNA detection in peripheral blood of normal people, benign breast disease patients and breast cancer patients, so as to act as the new techniques or indicators of early screening of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained and documented according to the local regulatory requirements prior to beginning specific protocol procedures.
* Age of at least 18 and at most 70 years.
* Normal people who works as the volunteers.
* Benign breast disease patients should be diagnosed with confirmed pathology after surgery.
* Breast cancer patients should be diagnosed with confirmed pathology after surgery, and with no clinical evidence of local recurrence or distant metastases. Complete staging work-up within 3 months prior to registration, which should be earlier than TNM IIA stage.
* Adequate organ function including normal red and white blood count, platelets, serum creatinine, bilirubin, and transaminases within normal range of the institution.

Exclusion Criteria:

* Known hypersensitivity reaction to the investigational compounds or incorporated substances.
* Local recurrence and/or metastasis of breast cancer.
* Pregnant or lactating patients. Patients of childbearing potential must have a negative pregnancy test (urine or serum) within 14 days prior to registration.
* Prior or concomitant secondary malignancy (except non-melanomatous skin cancer or carcinoma in situ of the uterine cervix).
* Other serious illness or medical condition that may interfere with the understanding and giving of informed consent and the conduct of the study.
* Concurrent treatment with other experimental drugs or any other anti-cancer therapy.
* Males.

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Three groups: normal people, benign breast disease patients and breast cancer patients in early stage.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
ctDNA test model for early screening of breast cancer | 2 years